CLINICAL TRIAL: NCT03248635
Title: Online Questionnaire Pre-Test Study
Brief Title: Questionnaire Pre-Test Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917139; 17-C-N139
Record Dates: First submitted 2017-08-11; First posted 2017-08-14 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Cancer
Keywords: Survey; Pre-Test
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Focus group: Male and female adults age 40-75

SUMMARY:
Background:

The Division of Cancer Epidemiology and Genetics does research into the causes of cancer and ways to prevent it. It uses data from questionnaires. Sometimes, pre-testing a questionnaire with a group of volunteers can help researchers find errors in it and learn ways to improve it.

Objectives:

To test a questionnaire for problems that might cause response errors and to develop ideas for improving it. To test how long it takes people to complete it.

Eligibility:

Adults ages 35-75. Volunteers both with and without a history of tobacco use and with or without a family history of cancer are needed.

Design:

Participants will be screened with a phone call.

Participants will be told what background data to bring to the 1 study visit.

An interviewer will give the participants the questionnaire. It will be done with pen and paper. It will take about 1 hour.

There will be multiple-choice and open-ended questions. They will be about lifestyle, medical, and environmental factors. Some of the questions will be about possibly illegal or highly sensitive behaviors.

Participants will note any questions that they find hard to answer for any reason. They will be asked to answer the best they can, but they can skip any question that they prefer not to answer.

The personal data of participants will be deleted when the study is done.

The interviewer will observe participants while they do the questionnaire. He or she will look for things like long pauses and confusion.

Participants will discuss the exam with the interviewer after they finish. This will take about 1 hour.

DETAILED DESCRIPTION:
The mission of the Division of Cancer Epidemiology and Genetics (DCEG) is to conduct broadbased, high quality, high impact research to uncover the causes of cancer and the means of its prevention. To this end, DCEG relies on epidemiologic data captured on self-reported questionnaires. The purpose of this pre-test study is to pilot a questionnaire to: (1) detect problems that might contribute to response errors; (2) develop ideas for improving the questionnaire in order to minimize such errors; and (3) assess the length of time to complete the questionnaire. If there are specific sections of the questionnaire that are skipped by all 30 initial participants, then six (6) additional, separate individuals may be invited to pre-test the questionnaire for sections that were missed by the initial set of participants. After a post-revision of the questionnaire based on the pre-test results, up to 10 additional, separate individuals will be invited to test the revised questionnaire for duration and comprehensibility.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Age 35 to 75
* Men or women
* Fluent in English
* Able to come to the SSS Durham, NC offices for the in-person interview
* Able to provide informed consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Convenience sample of adult volunteers in geographic proximity to contractor in Durham, NC
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Understanding of the Questionnaire | Time of Interview
  Response errors and comments on interpretation of questions and response categories, and the duration needed to complete the questionnaire modules.

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Purdue, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Social & Scientific Systems, INC, Durham, North Carolina, United States